CLINICAL TRIAL: NCT05652491
Title: The Role of Gut Microbiome in Predicting Comorbidities and Complications in Children With Inflammatory Bowel Disease
Status: Withdrawn | Type: Observational
Why Stopped: NIH Intramural Program is not the Responsible Party for this study and thus not responsible for registration.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000909; 000909-I
Record Dates: First submitted 2022-12-13; First posted 2022-12-15 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Pediatrics; Crohn's Disease; Ulcerative Colitis; Microbiota; Host-Microbiome Response; Natural History
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Subjects who are not diagnosed with IBD
- IBD Patients: New onset, treatment-naive pediatric IBD patients

SUMMARY:
Background:

Bacteria and other microorganisms that live in the intestines (the gut microbiome) play an important role in a person s health. The gut microbiome helps to regulate the immune system and control inflammation. Imbalances in the gut microbiome have been linked to illnesses such as inflammatory bowel disease (IBD). People diagnosed with IBD can have serious health problems. Researchers want to know more about how the gut microbiome affects the development and progression of IBD in children. In this natural history study, they will compare the gut microbiomes of healthy children with those who have IBD.

Objective:

To collect stool and samples of intestine tissue from children with and without IBD undergoing colonoscopy.

Eligibility:

People under 21 years old who are having a colonoscopy at the Inova Health System or Pediatric Specialists of Virginia.

Design:

Participants will fill out a questionnaire. They will answer questions about their history. Topics may include how they were fed as infants; how they were born; and how often they took antibiotics.

Stool and tissue samples from the intestines will be taken during the participants colonoscopy. They may also give samples of blood and urine.

Participants may be asked to provide additional stool, blood, and urine samples. They may do this up to 3 times per year. These samples may be collected at the clinic; they may also be collected at home and mailed to the researchers.

If they have more colonoscopies, participants may be asked for more tissue samples.

Participants will be enrolled for up to 10 years.

...

DETAILED DESCRIPTION:
The gut microbiome (community of microorganisms in the intestines) serves many important roles in healthy people, including immune system regulation and anti-inflammatory functions. A dysbiosis (imbalance) in the gut microbiome is associated with many immune mediated diseases, including inflammatory bowel disease (IBD). The microbiome is thought to play a central role in the development and propagation in IBD. Studies have shown that in IBD, the gut microbiome demonstrates increased pro-inflammatory bacteria, a reduction in anti-inflammatory bacteria and overall reduced diversity. Inflammatory bowel disease is complicated and comes at a high burden to those affected. While affecting both children and adults, patients diagnosed before 18 years of age often have more severe phenotypes than those diagnosed in adulthood. Patients affected by IBD often have many complications such as linear growth failure, decreased bone mineral indices, delayed puberty, malnutrition and need for surgeries. At this time, we have limited ability to predict which patients will go on to develop complications and the time points in which these may occur.

Further, there are many comorbidities present in patients with IBD including dermatologic manifestations, hepatobiliary disease, other immune-mediated disease such as celiac disease as well as endocrinopathies. Children with IBD and these comorbid conditions are thought to have higher morbidity and decreased quality of life. While the gut microbiome is thought to mediate the development of many of these diseases, there is little literature associating clinical and microbiome drivers of those with IBD and these additional comorbidities.

Given that the microbiome may have a role in potentiating the inflammatory pathways contributing to IBD, there is potential to identify microbial signatures to help determine disease outcomes such as complications and response to treatment. In this study, we intend to examine differences in the microbiome diversity and composition in children with IBD and controls. We will then follow subjects longitudinally to determine initial microbiota signatures and changes for those who develop comorbidities, complications and therapy responsiveness.

We hope that by elucidating the microbiome of these children, we will have the opportunity to better understand the pathogeneses of co-morbid diseases, ultimately enabling the development of microbiome-based therapeutics for these conditions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients 0<=21 years of age undergoing colonoscopy will be approached for enrollment in this study.

EXCLUSION CRITERIA:

Participants carrying known diagnosis of IBD, including Crohn's disease, Ulcerative Colitis or IBD-Unspecified. However, patients with IBD suspected prior to colonoscopy can be included.

Max Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients already planned to have a colonoscopy as per their primary gastroenterologist seen at Pediatric Specialists of Virginia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
differences in fecal/intestinal microbiome | at diagnosis
  Determine differences in fecal/intestinal microbiome of patients IBD as compared to controls
differences in fecal microbiome diversity and composition | longitudinal throughout follow up
  Determine differences in fecal microbiome diversity and composition in children with IBD with and without comorbidities
microbiome signatures for newly diagnosed IBD patients | longitudinal throughout follow up
  Determine if microbiome signatures for newly diagnosed IBD patients can predict complications and response to treatments

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra K Hourigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland
  - Inova Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
.Raw, de-identified data may be shared as part of publication. This will only be sequencing data, any other data will be compiled.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Exact time frame is unknown. Will be completed as part of publication requirements.
Access Criteria: Raw, de-identified data may be shared as part of publication. This will only be sequencing data, any other data will be compiled. No other current plans for sharing data exist.